CLINICAL TRIAL: NCT02512744
Title: Reducing Decannulation Time in Critically-ill Tracheostomized Patients: Decannulation Capping Trial Protocol vs Frequency Aspiration Protocol (REDECAP)
Brief Title: Reducing Decannulation Time: Limitation of Decannulation Capping Trials (REDECAP)
Acronym: REDECAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Virgen de la Salud (Other)
Responsible Party: Principal Investigator, Gonzalo Hernandez Martinez, MD, Hospital Virgen de la Salud
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3/7/2015 n67
Record Dates: First submitted 2015-07-27; First posted 2015-07-31 (Estimated); Last update posted 2018-08-07 (Actual); Status verified 2018-08

CONDITIONS: Tracheostomy; Airway Management; Respiratory Therapy
Keywords: Tracheostomy; Decannulation; Adult airway management

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Capping trial protocol (No Intervention): Decannulation protocol based on tolerance to 24 hours capping trial to decide when to decannulate.
  Decapping during the capping trial for aspiration of respiratory secretions is considered a failure criteria of the trial.
  High flow conditioned oxygen therapy through tracheal cannula will be applied during periods out of capping trials.
- Suctioning frequency protocol (Experimental): Decannulation protocol based on suctioning frequency to decide when to decannulate (criteria: ≤2 aspirations every 8 h along 24 consecutive hours).
  Intervention: suctioning frequency of respiratory secretions will be recorded untill fulfill decannulation criteria. Capping trials will not be allowed in this group.
  High flow conditioned oxygen therapy will be applied through tracheal cannula during all the study period.
  Interventions: Procedure: Decannulation protocol.; Device: High flow conditioned oxygen therapy

INTERVENTIONS:
Procedure: Decannulation protocol. — Comparison of two different decannulation protocols: one protocol based on capping trial tolerance to decide when to decannulate vs. protocol based on suctioning frequency of respiratory secretions to decide when to decannulate (criteria: ≤2 aspirations every 8 h along 24 consecutive hours).
  Arms: Suctioning frequency protocol
Device: High flow conditioned oxygen therapy — High flow conditioned oxygen therapy will be applied during all study period through tracheal cannula in the experimental arm (suctioning frequency based protocol) and during periods out of capping trials in the control arm (capping trials based protocol).
  Other Names: OptiflowTM, Fisher&Paykel, Auckland, New Zealand.
  Arms: Suctioning frequency protocol

SUMMARY:
Multicenter randomized trial centered on critically-ill tracheostomized patients, comparing two different decannulation protocols:

1. based on capping trials to decide decannulation,
2. based on the aspiration frequency to decide decannulation time. High-flow conditioned oxygen therapy will be applied to all patients through the tracheal cannula. In patients included in the suctioning frequency based protocol along the study period and in patients included in the capping trial protocol along periods out of capping trials.

ELIGIBILITY:
Inclusion Criteria:

* Critically-ill tracheostomized patients weaned from mechanical ventilation (24 consecutive hours disconnected).

Exclusion Criteria:

* Patients consedered non-decannulable at time of randomization:

  1. unconscious patient (motor component of GCS score <6 points).
  2. Severe swallowing function (based on drink test).
  3. Airway patency problem (based of intolerance of occlusion test).
  4. Neuromuscular diseases.
  5. Patients with a Sabadell score >2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
Decannulation time | Patients will be followed for the duration of hospital stay, an expected average of 3 months
  Time since weaning from mechanical ventilation (24 consecutive hours disconnected) to decannulation

SECONDARY OUTCOMES:
Decannulation failure | Patients will be followed for the duration of hospital stay, an expected average of 3 months
  Number of patients requiring recannulation during hospital stay / number of patients included in the group X 100
Intensive Care Unit Lenght of stay | Patients will be followed for the duration of ICU stay, an expected average of 2 months
  Time since ICU admission to ICU discharge
Hospital lenght of stay | Patients will be followed for the duration of hospital stay, an expected average of 3 months
  Time since hospital admission to hospital discharge
ICU mortality | Patients will be followed for the duration of ICU stay, an expected average of 2 months
  ICU mortality in every study group
Hospital mortality | Patients will be followed for the duration of hospital stay, an expected average of 3 months
  Hospital mortality in every study group
Respiratory infection | Patients will be followed for the duration of hospital stay, an expected average of 3 months
  Post-randomization pneumonia and tracheobronchitis rate in every study group

CONTACTS AND LOCATIONS:
Overall Officials: GONZALO HERNANDEZ, MD, Study Chair — Hospital Virgen de la Salud
Locations (5):
- Spain (5):
  - Hospital Del Mar, Barcelona
  - Hospital Universitario Vall D´Ebron, Barcelona
  - Hospital Universitario de Ciudad Real, Ciudad Real
  - Hospital Universitario Ramon Y Cajal, Madrid
  - Hospital Virgen de La Salud, Toledo

REFERENCES:
- [Derived] Hernandez Martinez G, Rodriguez ML, Vaquero MC, Ortiz R, Masclans JR, Roca O, Colinas L, de Pablo R, Espinosa MD, Garcia-de-Acilu M, Climent C, Cuena-Boy R. High-Flow Oxygen with Capping or Suctioning for Tracheostomy Decannulation. N Engl J Med. 2020 Sep 10;383(11):1009-1017. doi: 10.1056/NEJMoa2010834. PMID 32905673